CLINICAL TRIAL: NCT01592747
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study of the Safety and Efficacy of Memantine in Pediatric Patients With Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS) Previously Treated With Memantine
Brief Title: Withdrawal Study of Memantine in Pediatric Patients With Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified Previously Treated With Memantine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEM-MD-68
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-03

CONDITIONS: Autistic Disorder; Autism; Asperger's Disorder; Asperger Syndrome; Autism Spectrum Disorders; Pervasive Developmental Disorder - Not Otherwise Specified (PDD-NOS)
Keywords: Asperger's; Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS); Memantine; Pediatric Disorder; Randomized Controlled Trial
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Autism Spectrum Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Memantine 1 (Experimental): Patients randomized to the full dose arm will continue taking memantine at the same tolerability and weight-based dose achieved in lead-in Study MEM-MD-91. Dosing will be once daily for up to 12 weeks.
  Interventions: Drug: Memantine Hydrochloride (HCl)
- Memantine 2 (Experimental): Patients randomized to the reduced dose arm will take memantine at the tolerability and weight based dose that they received in lead in Study MEM-MD-91 reduced by at least 50%. Dosing will be once daily for up to 12 weeks.
  Interventions: Drug: Memantine Hydrochloride (HCl)
- Placebo (Placebo Comparator): Dosing will be once daily for up to 12 weeks.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Memantine Hydrochloride (HCl) — Extended Release Dose ranging from 3-15mg/day; administered orally
  Arms: Memantine 1
Drug: Memantine Hydrochloride (HCl) — Extended Release Dose ranging from 3mg every other day to 6mg/day; administered orally.
  Arms: Memantine 2
Drug: Placebo capsules — Once daily, oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this randomized withdrawal study is to evaluate the safety, tolerability, and efficacy of memantine compared with placebo in pediatric patients with autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS).

DETAILED DESCRIPTION:
This clinical study was a 12-week, multicenter, double-blind, placebo-controlled, randomized withdrawal study in pediatric outpatients with autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS). Patients who completed at least 12 weeks of study drug exposure and met protocol specified responder criterion in lead in Study MEM-MD-91 (NCT01592786) at two consecutive visits separated by at least two weeks were eligible to transition to this study. The responder criterion was defined as having at least a 10 point improvement (reduction in score) in the Social Responsiveness Scale (SRS) total raw score relative to the Visit 1 total raw score in Study MEM-MD-91.

Weight based dose limits were selected in this study to ensure that exposure in terms of area under the curve (AUC) was less than the predefined limit of 2100 ng·h/mL which represents a 10-fold lower exposure than observed at the NOAEL(No observed adverse effect level) of 15 mg/kg/day in juvenile rats.

The weight-based dose limits in this study were as follows:

* Group A: ≥ 60 kg; maximum 15 mg/day
* Group B: 40-59 kg; maximum 9 mg/day
* Group C: 20-39 kg; maximum 6 mg/day
* Group D: < 20 kg; maximum 3 mg/day

ELIGIBILITY:
Inclusion Criteria:

1. Completed at least 12 weeks of exposure to study drug in lead-in study MEM-MD-91 (NCT01592786)
2. Met responder criterion at two consecutive visits separated by at least two weeks in lead-in study MEM-MD-91
3. Provide written informed assent, when developmentally appropriate, to participate in the study before conduct of any study-specific procedures. The parent/guardian/LAR must provide written informed consent before the patient's participation in the study. A separate written informed consent for the caregiver must also be obtained before the conduct of any study specific procedures
4. Have a knowledgeable caregiver who is capable of providing reliable information about the patient's condition, attending all clinic visits with the patient, and overseeing the administration of study drug. Every effort should be made to maintain the same caregiver as used in the lead-in study throughout this study
5. Have normal results from the physical examination, laboratory tests, ECG, and vital signs at Visit 1 of this study (last visit of Study MEM-MD-91). Any abnormal findings must be deemed not clinically significant by the Investigator and documented
6. Be able to speak and understand English sufficiently (or their native language if this can be accommodated by the site), as well as have a caregiver and parent/guardian/LAR who is able to speak and understand English sufficiently (or their native language if this can be accommodated by the site), to comprehend the nature of the study and to allow for the completion of all study assessments
7. Have a family that is sufficiently organized and stable to guarantee adequate safety monitoring and continuous attendance to clinic visits for the duration of the study
8. Females who are 9 years and older or who have had onset of menses must have a negative urine pregnancy test at Visit 1
9. Age of 6 years to 12 years at the time of entry into lead in study MEM-MD-91

Exclusion Criteria:

1. Patients with a concurrent medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger the patient's well being
2. Significant risk of suicidality based on the Investigator's judgment, the Aberrant Behavior Checklist-Irritability subscale (ABC-I), or if appropriate, as indicated by a response of "yes" to questions 4 or 5 in the suicidal ideation section of the Children's C-SSRS (Columbia-Suicide Severity Rating Scale) or any suicidal behavior.
3. Patients with evidence or history of malignancy (other than excised basal cell carcinoma) or any significant hematologic, endocrine, cardiovascular (including any rhythm disorder), neurologic, respiratory, renal, hepatic, or gastrointestinal disease
4. Female patients of child-bearing potential who are not using or not willing to use a conventional method of contraception approved by the PI. Abstinence is an acceptable method of contraception
5. Patients requiring treatment with prohibited concomitant medications
6. Patients who, in the opinion of the Investigator, might not be suitable for the study
7. Employee or immediate relative of an employee of Forest Laboratories, Inc., any of its affiliates or partners, or the study center

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 479 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lateiner, MS, MBA, Study Director — Forest Research Institute, Inc.- A Subsidiary of Forest Laboratories, Inc.
Locations (94):
- United States (64):
  - Forest Investigative Site 068, Dothan, Alabama
  - Forest Investigative Site 005, Phoenix, Arizona
  - Forest Investigative Site 055, Tucson, Arizona
  - Forest Investigative Site 077, Little Rock, Arkansas
  - Forest Investigative Site 054, Glendale, California
  - Forest Investigative Site 109, Imperial, California
  - Forest Investigative Site 096, Los Angeles, California
  - Forest Investigative Site 021, San Francisco, California
  - Forest Investigative Site 026, Santa Ana, California
  - Forest Investigative Site 002, Stanford, California
  - Forest Investigative Site 078, Boulder, Colorado
  - Forest Investigative Site 073, Centennial, Colorado
  - Forest Investigative Site 052, Washington D.C., District of Columbia
  - Forest Investigative Site 075, Bradenton, Florida
  - Forest Investigative Site 080, Gainesville, Florida
  - Forest Investigative Site 117, Jacksonville, Florida
  - Forest Investigative Site 065, Maitland, Florida
  - Forest Investigative Site 118, Miami, Florida
  - Forest Investigative Site 085, Oakland Park, Florida
  - Forest Investigative Site 115, Orange City, Florida
  - Forest Investigative Site 125, Orlando, Florida
  - Forest Investigative Site 062, Orlando, Florida
  - Forest Investigative Site 067, Tampa, Florida
  - Forest Investigative Site 101, Wellington, Florida
  - Forest Investigative Site 102, Libertyville, Illinois
  - Forest Investigative Site 023, Naperville, Illinois
  - Forest Investigative Site 082, Evansville, Indiana
  - Forest Investigative Site 056, Indianapolis, Indiana
  - Forest Investigative Site 106, Wichita, Kansas
  - Forest Investigative Site 061, Louisville, Kentucky
  - Forest Investigative Site 095, Lake Charles, Louisiana
  - Forest Investigative Site 086, Rockville, Maryland
  - Forest Investigative Site 059, Newton, Massachusetts
  - Forest Investigative Site 108, Springfield, Massachusetts
  - Forest Investigative Site 116, Lincoln, Nebraska
  - Forest Investigative Site 097, Lincoln, Nebraska
  - Forest Investigative Site 130, Henderson, Nevada
  - Forest Investigative Site 104, Las Vegas, Nevada
  - Forest Investigative Site 136, Neptune City, New Jersey
  - Forest Investigative Site 127, Toms River, New Jersey
  - Forest Investigative Site 081, Albuquerque, New Mexico
  - Forest Investigative Site 107, Albuquerque, New Mexico
  - Forest Investigative Site 072, Chapel Hill, North Carolina
  - Forest Investigative Site 069, Avon Lake, Ohio
  - Forest Investigative Site 001, Columbus, Ohio
  - Forest Investigative Site 019, Oklahoma City, Oklahoma
  - Forest Investigative Site 092, Tulsa, Oklahoma
  - Forest Investigative Site 053, Gresham, Oregon
  - Forest Investigative Site 132, Johnstown, Pennsylvania
  - Forest Investigative Site 131, McMurray, Pennsylvania
  - Forest Investigative Site 100, Media, Pennsylvania
  - Forest Investigative Site 105, Charleston, South Carolina
  - Forest Investigative Site 090, Memphis, Tennessee
  - Forest Investigative Site 057, Nashville, Tennessee
  - Forest Investigative Site 051, Houston, Texas
  - Forest Investigative Site 070, The Woodlands, Texas
  - Forest Investigative Site 028, Clinton, Utah
  - Forest Investigative Site 141, Ogden, Utah
  - Forest Investigative Site 029, Salt Lake City, Utah
  - Forest Investigative Site 064, Charlottesville, Virginia
  - Forest Investigative Site 113, Norfolk, Virginia
  - Forest Investigative Site 071, Bothell, Washington
  - Forest Investigative Site 119, Charleston, West Virginia
  - Forest Investigative Site 063, Middleton, Wisconsin
- Belgium (2):
  - Forest Investigative Site 204, Brussels
  - Forest Investigative Site 203, Brussels
- Colombia (2):
  - Forest Investigative Site 228, Bello
  - Forest Investigative Site 226, Bogotá
- Forest Investigative Site 276, Tallinn, Estonia
- Forest Investigative Site 329, Bron, France
- Hungary (3):
  - Forest Investigative Site 381, Budapest
  - Forest Investigative Site 376, Budapest
  - Forest Investigative Site 378, Budapest
- Forest Investigative Site 401, Kopavogur, Iceland
- Italy (2):
  - Forest Investigative Site 453, Roma
  - Forest Investigative Site 452, Siena
- Forest Investigative Site 526, Wellington, New Zealand
- Poland (4):
  - Forest Investigative Site 579, Gdansk
  - Forest Investigative Site 578, Gdansk
  - Forest Investigative Site 576, Kobierzyce
  - Forest Investigative Site 577, Warsaw
- Serbia (4):
  - Forest Investigative Site 626, Belgrade
  - Forest Investigative Site 627, Belgrade
  - Forest Investigative Site 629, Niš
  - Forest Investigative Site 628, Novi Sad
- Forest Investigative Site 676, Cape Town, Western Cape, South Africa
- South Korea (4):
  - Forest Investigative Site 704, Yangsan, Gyeongsangnam-do
  - Forest Investigative Site 702, Seoul
  - Forest Investigative Site 703, Seoul
  - Forest Investigative Site 701, Seoul
- Forest Investigative Site 728, Sabadell, Barcelona, Spain
- Ukraine (3):
  - Forest Investigative Site 807, Kharkiv
  - Forest Investigative Site 802, Kherson,Vil. Stepanivka
  - Forest Investigative Site 804, Kyiv

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a ten month period, from September of 2012 to June of 2013, at 92 study sites, located in the Untied States and 14 other countries.
Pre-assignment Details: Patients who completed at least 12 weeks of exposure to open-label memantine and met the responder criterion at 2 consecutive visits separated by at least 2 weeks during lead-in study MEM-MD-91 were eligible to enroll into this study.
Groups:
- Placebo: Dose-matched placebo, oral administration, once per day.
- Memantine Reduced Dose: Memantine, 3mg every other day, 3mg per day, or 6mg per day depending on weight group and tolerability. Oral administration once per day.
- Memantine Full-Dose: Memantine, 3mg, 6mg, 9mg, 12mg or 15mg, depending on weight group and tolerability. Oral administration, once per day.
Period: Overall Study
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Started | 160 (Based on Randomized Population) | 161 (Based on Randomized Population) | 158 (Based on Randomized Population)
Completed | 44 | 50 | 50
Not Completed | 116 | 111 | 108
Not completed — Loss of Therapeutic Response | 107 | 108 | 100
Not completed — Inclusion/Exclusion criteria not met | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 4
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Other Reasons | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 479 patients were screened and randomized. Of these, 477 patients received at least 1 dose of double-blind investigational product (Safety Population). The baseline characteristics presented here are for the Safety population.
Groups:
- Memantine Full-Dose: Memantine, 3mg, 6mg, 9mg, 12mg or 15mg depending on weight group and tolerability. Oral administration, once per day.
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose | Total
Number analyzed (Participants) | 160 | 160 | 157 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.9 (2.0) | 9.2 (1.9) | 9.2 (1.9) | 9.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 28 | 25 | 71
  Male | 142 | 132 | 132 | 406
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 22 | 15 | 60
  Not Hispanic or Latino | 137 | 138 | 142 | 417
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 138 | 141 | 140 | 419
  Black or African American | 10 | 9 | 7 | 26
  Asian | 7 | 5 | 8 | 20
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Other | 4 | 3 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 134 | 125 | 126 | 385
  Belgium | 2 | 1 | 1 | 4
  Colombia | 1 | 2 | 2 | 5
  Estonia | 0 | 1 | 0 | 1
  France | 1 | 4 | 2 | 7
  Hungary | 3 | 3 | 2 | 8
  Iceland | 0 | 3 | 0 | 3
  Italy | 2 | 1 | 1 | 4
  Korea, Republic of | 6 | 3 | 5 | 14
  New Zealand | 0 | 1 | 1 | 2
  Poland | 5 | 6 | 10 | 21
  Serbia | 3 | 6 | 5 | 14
  South Africa | 0 | 0 | 1 | 1
  Spain | 1 | 0 | 1 | 2
  Ukraine | 2 | 4 | 0 | 6
Autism Spectrum Disorder Subtype [Count of Participants; unit: Participants]
  Autism | 101 | 99 | 100 | 300
  Asperger's Disorder | 30 | 30 | 27 | 87
  PDD-NOS | 29 | 31 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Meeting the Criterion for Loss of Therapeutic Response (LTR) by the End of the Study (Based on Observed Cases)
Description: Loss of Therapeutic response is defined as a worsening (increase) of at least 10 points in Social Responsiveness Scale (SRS) total raw score relative to the Visit 1 (randomization) score. The Social Responsiveness Scale (SRS) is a 65-item informant-rated assessment with total raw score ranging from 0 (no impairment) to 195 (severe social impairment). Each item is associated with 1 of 5 subscales (social awareness, social cognition, social communication, social motivation and autistic mannerisms). Each item is rated on a 4-point scale from 1 (not true) to 4 (almost always true). The scores are then transposed to a scale from 0 to 3 and scores are summed within each of the 5 subscales. A higher score indicates greater severity of social impairment.
Time Frame: Baseline (Visit 1) to week 12
Population: All efficacy analyses were based on the Intent-to-treat (ITT) Population. Of the 479 randomized patients, 471 patients were in the ITT Population (ie, had at least 1 dose of double-blind investigational product and at least 1 assessment of the Social Responsiveness Scale (SRS) total raw score during the double-blind treatment period.)
Measure: Number; unit: Percentage of patients with LTR
Groups:
- Memantine Reduced Dose: Memantine, 3mg every other day, 3mg per day, or 6mg per day depending on weight group and tolerability. Oral administration, once per day.
- Memantine Full-Dose: Memantine, 3mg, 6mg, 9mg, 12mg or 15mg; oral administration. Once per day.
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 158 | 160 | 153
Percentage of patients with LTR | 69.0 | 67.5 | 66.7
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Cochran-Mantel-Haenszel test was performed controlling for Autism Spectrum Disorder (ASD) subtype. Odds ratio was calculated for placebo vs. memantine full dose; Test type: Superiority or Other; p = 0.6590, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.8]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Cochran-Mantel-Haenszel test was performed controlling for Autism Spectrum Disorder (ASD) subtype. Odds ratio was calculated for placebo vs. Memantine reduced dose; Test type: Superiority or Other; p = 0.7839, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.7]

2. Secondary Outcome: Time to First Loss of Therapeutic (LTR) Response
Description: Time to the first visit when a patient shows LTR following randomization to memantine or placebo.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 158 | 160 | 153
Days | 29 [28 to 42] | 33 [28 to 56] | 30 [28 to 44]

3. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Speech Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Speech Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: Of the 479 randomized patients, 471 patients were included in the Intent to Treat (ITT) Population. Within the ITT population, 466 patients had post-baseline assessment of the Children's Communication Checklist-2 (CCC-2).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.1 (0.2) | 0.1 (0.2) | 0.2 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.8136, ANCOVA; Least squares mean difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.9244, ANCOVA; Least squares mean difference = -0.0, 95% CI 2-sided [-0.6 to 0.5]

4. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Syntax Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Syntax Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.0 (0.2) | 0.3 (0.2) | 0.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.7611, ANCOVA; Least squares mean difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.3176, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.3 to 0.9]

5. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Semantics Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Semantics Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.3 (0.2) | 0.7 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.9020, ANCOVA; Least squares mean difference = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.1279, ANCOVA; Least squares mean difference = 0.4, 95% CI 2-sided [-0.1 to 1.0]

6. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Coherence Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Coherence Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.7 (0.3) | 1.0 (0.3) | 1.0 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.4144, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 1.1]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.4212, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 1.0]

7. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Initiation Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Initiation Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 1.4 (0.3) | 1.6 (0.3) | 1.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.6238, ANCOVA; Least squares mean difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.5957, ANCOVA; Least squares mean difference = 0.2, 95% CI 2-sided [-0.5 to 0.9]

8. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Scripted Language Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Scripted language Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.8 (0.2) | 1.1 (0.2) | 0.9 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.8640, ANCOVA; Least squares mean difference = 0.1, 95% CI 2-sided [-0.6 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.4362, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 0.9]

9. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Context Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Context Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.9 (0.3) | 0.8 (0.3) | 0.8 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.7182, ANCOVA; Least squares mean difference = -0.1, 95% CI 2-sided [-0.8 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.8390, ANCOVA; Least squares mean difference = -0.1, 95% CI 2-sided [-0.8 to 0.6]

10. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Nonverbal Communication Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Nonverbal communication Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 1.2 (0.3) | 1.5 (0.3) | 1.8 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.0813, ANCOVA; Least squares mean difference = 0.7, 95% CI 2-sided [-0.1 to 1.4]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.4365, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 1.0]

11. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Social Relations Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Social Relations Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 1.5 (0.3) | 1.8 (0.3) | 1.8 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.4213, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.4267, ANCOVA; Least squares mean difference = 0.3, 95% CI 2-sided [-0.4 to 1.0]

12. Secondary Outcome: Change From Baseline in Children's Communication Checklist-2 (CCC-2) - Interests Subscale at Week 12
Description: The Children's Communication Checklist-2 (CCC-2) is a validated, norm-referenced, informant-rated scale that evaluates difficulties (items 1-50) and strengths (items 51-70) in communication. There are 10 sub-scales consisting of 7 items each. The Children's Communication Checklist-2 (CCC-2) Interests Subscale consists of 7 items rated from 0 (less than once a week or never) to 3 (several times [more than twice] a day or always), with a total raw score of 0 (mildest) to 21 (most severe).
Time Frame: Baseline (Visit 1) to week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Number analyzed (Participants) | 154 | 159 | 153
units on a scale | 0.9 (0.3) | 1.3 (0.3) | 1.2 (0.3)
Statistical Analysis 1: Comparison: Placebo vs Memantine Full-Dose; Test type: Superiority or Other; p = 0.3713, ANCOVA; Least squares mean difference = 0.3, 95% CI [-0.4 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs Memantine Reduced Dose; Test type: Superiority or Other; p = 0.2855, ANCOVA; Least squares mean difference = 0.4, 95% CI 2-sided [-0.3 to 1.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a 14 month period from September of 2012 to October of 2013 at 92 study centers in the United States and 14 other countries.
Description: Safety results are based on Safety Population (ie, all randomized patients who took at least 1 dose of double-blind study drug).
Groups:
- Memantine Reduced Dose: Memantine, 3mg every other day, 3mg per day, or 6mg per day. Oral administration.
Arm/Group | Placebo | Memantine Reduced Dose | Memantine Full-Dose
Serious Adverse Events (participants affected / at risk) | 0/160 | 1/160 | 0/157
Other Adverse Events (participants affected / at risk) | 8/160 | 5/160 | 4/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Memantine Reduced Dose (N=160) | Memantine Full-Dose (N=157)
Furuncle (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=160) | Memantine Reduced Dose (N=160) | Memantine Full-Dose (N=157)
Irritability (General disorders) | 8 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.